CLINICAL TRIAL: NCT03356964
Title: Impact of Step-down Approach During Late Follicular Phase in Recombinant FSH-stimulation Dosage for IVF on Progesterone Level on the Day of Final Oocyte Maturation
Brief Title: Step Down FSH Approach and Late Follicular Phase in Progesterone Level
Acronym: FSH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Prof Dr. Human Fatemi, Professor Doctor, ART Fertility Clinics LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1612-ABU-084-HF
Record Dates: First submitted 2017-11-14; First posted 2017-11-29 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Progesterone Resistance
Keywords: endometrial receptivity progesterone elevation
MeSH Terms: conditions — Progesterone Resistance | interventions — Follicle Stimulating Hormone; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Follicle stimulating Hormone will be applied, starting from day 3 of the cycle, the dosage will be choosen between Gonal F 150 - 225 IU, according to the ovarian reserve parameters (13). The stimulation dosage will remain unchanged until the criteria for final oocyte maturation are met (≥ 3 follicles of ≥ 17 mm).
  Interventions: Drug: follicle stimulating hormone
- Study group (Experimental): Follicle stimulating Hormone will be applied, starting from day 3 of the cycle, the dosage will be choosen between Gonal F 150 - 225 IU, according to the ovarian reserve parameters (LaMarca et al.). As soon as ≥ 3 follicle of a size of 14mm are seen, the stimulation dosage will be reduced daily by 12.5 IU recFSH until the criteria for final oocyte maturation are met (≥ 3 follicles of ≥ 17 mm).
  Interventions: Drug: follicle stimulating hormone

INTERVENTIONS:
Drug: follicle stimulating hormone — Follicle stimulating hormone( will be chosen according to ovarian reserve parameters in the study group the dosage will be reduced in the control group it will remain unchanged
  Other Names: Gonal-F

SUMMARY:
Step-down approach and late follicular phase progesterone level

DETAILED DESCRIPTION:
The study will be performed using the stimulation medication Gonal-F which is a recombinant FSH-preparation. Due to application as pen-device, it allows reduction of the stimulation dosage in steps of 12.5IU.

It is important to evaluate the dynamics of progesterone-rise after final oocyte maturation, as this dynamic might also have an influence on the receptivity of the endometrium.

ELIGIBILITY:
Inclusion Criteria:

* Primary / secondary infertility with the indication for IVF/ICSI
* Patients age 18 - 40 years
* 60 kg up to and including 90 kg
* BMI of 18-32 kg/m2
* Menstrual cycle length of 24-35 days

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

Exclusion criteria:

* presence or history of an endocrine abnormality
* abnormal outcome of blood biochemistry or hematology
* relevant ovarian-, tubal- or uterine-pathology that could interfere with the ovarian stimulation treatment
* history of ovarian hyper-response (more than 30 follicles ≥ 11 mm) or ovarian hyper-stimulation syndrome (OHSS), polycystic ovary syndrome (PCOS)
* History of poor ovarian response, according to the Rotterdam-criteria (Ferrarretti et al.)
* ovarian reserve parameter, indicating the risk of poor ovarian response (AFC < 5 and AMH < 0,5ng/ml) (14)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female population who will undergo IVF treatment
Enrollment: 127 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Impact of dose reduction in recFSH for IVF on the progesterone level. | 1year and 6 months
  Whether higher progesterone levels on the day of trigger will lead to rapid rise of progesterone after ovulation induction compared to lower progesterone levels.

CONTACTS AND LOCATIONS:
Overall Officials: Human Fatemi, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- IVI Middle East Fertilty Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourgain C, Ubaldi F, Tavaniotou A, Smitz J, Van Steirteghem AC, Devroey P. Endometrial hormone receptors and proliferation index in the periovulatory phase of stimulated embryo transfer cycles in comparison with natural cycles and relation to clinical pregnancy outcome. Fertil Steril. 2002 Aug;78(2):237-44. doi: 10.1016/s0015-0282(02)03228-4. PMID 12137857
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Filicori M, Cognigni GE, Pocognoli P, Tabarelli C, Spettoli D, Taraborrelli S, Ciampaglia W. Modulation of folliculogenesis and steroidogenesis in women by graded menotrophin administration. Hum Reprod. 2002 Aug;17(8):2009-15. doi: 10.1093/humrep/17.8.2009. PMID 12151429
- [Background] Givens CR, Schriock ED, Dandekar PV, Martin MC. Elevated serum progesterone levels on the day of human chorionic gonadotropin administration do not predict outcome in assisted reproduction cycles. Fertil Steril. 1994 Nov;62(5):1011-7. doi: 10.1016/s0015-0282(16)57066-6. PMID 7926111
- [Background] Griesinger G, Mannaerts B, Andersen CY, Witjes H, Kolibianakis EM, Gordon K. Progesterone elevation does not compromise pregnancy rates in high responders: a pooled analysis of in vitro fertilization patients treated with recombinant follicle-stimulating hormone/gonadotropin-releasing hormone antagonist in six trials. Fertil Steril. 2013 Dec;100(6):1622-8.e1-3. doi: 10.1016/j.fertnstert.2013.08.045. Epub 2013 Sep 29. PMID 24083873
- [Background] Kyrou D, Al-Azemi M, Papanikolaou EG, Donoso P, Tziomalos K, Devroey P, Fatemi HM. The relationship of premature progesterone rise with serum estradiol levels and number of follicles in GnRH antagonist/recombinant FSH-stimulated cycles. Eur J Obstet Gynecol Reprod Biol. 2012 Jun;162(2):165-8. doi: 10.1016/j.ejogrb.2012.02.025. Epub 2012 Mar 17. PMID 22425288
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Lawrenz B, Beligotti F, Engelmann N, Gates D, Fatemi HM. Impact of gonadotropin type on progesterone elevation during ovarian stimulation in GnRH antagonist cycles. Hum Reprod. 2016 Nov;31(11):2554-2560. doi: 10.1093/humrep/dew213. Epub 2016 Sep 12. PMID 27619773
- [Background] Schoolcraft W, Sinton E, Schlenker T, Huynh D, Hamilton F, Meldrum DR. Lower pregnancy rate with premature luteinization during pituitary suppression with leuprolide acetate. Fertil Steril. 1991 Mar;55(3):563-6. PMID 1900481
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Embryo cryopreservation rescues cycles with premature luteinization. Fertil Steril. 2010 Feb;93(2):636-41. doi: 10.1016/j.fertnstert.2009.01.134. Epub 2009 Mar 17. PMID 19296941
- [Background] Ubaldi F, Smitz J, Wisanto A, Joris H, Schiettecatte J, Derde MP, Borkham E, Van Steirteghem A, Devroey P. Oocyte and embryo quality as well as pregnancy rate in intracytoplasmic sperm injection are not affected by high follicular phase serum progesterone. Hum Reprod. 1995 Dec;10(12):3091-6. doi: 10.1093/oxfordjournals.humrep.a135864. PMID 8822420
- [Background] Venetis CA, Kolibianakis EM, Papanikolaou E, Bontis J, Devroey P, Tarlatzis BC. Is progesterone elevation on the day of human chorionic gonadotrophin administration associated with the probability of pregnancy in in vitro fertilization? A systematic review and meta-analysis. Hum Reprod Update. 2007 Jul-Aug;13(4):343-55. doi: 10.1093/humupd/dmm007. Epub 2007 Apr 3. PMID 17405832
- [Background] Venetis CA, Kolibianakis EM, Bosdou JK, Tarlatzis BC. Progesterone elevation and probability of pregnancy after IVF: a systematic review and meta-analysis of over 60 000 cycles. Hum Reprod Update. 2013 Sep-Oct;19(5):433-57. doi: 10.1093/humupd/dmt014. Epub 2013 Jul 4. PMID 23827986
- [Background] Yding Andersen C, Bungum L, Nyboe Andersen A, Humaidan P. Preovulatory progesterone concentration associates significantly to follicle number and LH concentration but not to pregnancy rate. Reprod Biomed Online. 2011 Aug;23(2):187-95. doi: 10.1016/j.rbmo.2011.04.003. Epub 2011 Apr 28. PMID 21665546
- [Derived] Lawrenz B, Coughlan C, Melado L, Digma S, Sibal J, Jean A, Fatemi HM. Step-Down of FSH- Dosage During Ovarian Stimulation - Basic Lessons to Be Learnt From a Randomized Controlled Trial. Front Endocrinol (Lausanne). 2021 Apr 13;12:661707. doi: 10.3389/fendo.2021.661707. eCollection 2021. PMID 33927696